CLINICAL TRIAL: NCT00768482
Title: A Single Cross-Over, Open-Label Study of the Relative Bioavailability of Probuphine Versus Buprenorphine Sublingual Tablets at Steady State in Patients With Opioid Dependence
Brief Title: A Bioavailability and Safety Study of Probuphine Versus Sublingual Buprenorphine in Patients With Opioid Dependence
Acronym: PRO-810
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: This study was terminated for reasons not related to efficacy or safety
Sponsor: Titan Pharmaceuticals (Industry)
Responsible Party: Sponsor
Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PRO-810
Record Dates: First submitted 2008-10-07; First posted 2008-10-08 (Estimated); Last update posted 2018-12-31 (Actual); Status verified 2017-06

CONDITIONS: Opioid Dependence
Keywords: opioid dependence; opioid addiction; buprenorphine; methadone; heroin; implant; opioid withdrawal; opioid pain medication; suboxone
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Probuphine (Experimental): Patients are first inducted on SL BPN, and then switched to 4 Probuphine implants
  Interventions: Drug: Probuphine (buprenorphine implant); Drug: Sublingual Buprenorphine

INTERVENTIONS:
Drug: Probuphine (buprenorphine implant) — Implantable formulation of buprenorphine made of buprenorphine HCl/ethylene vinyl acetate, considered a drug. (4 implants)
Drug: Sublingual Buprenorphine — 16 mg/day, QD

SUMMARY:
This study will measure the amount of buprenorphine found in the blood after taking sublingual buprenorphine tablets versus after implantation with 4 Probuphine (buprenorphine implants).

DETAILED DESCRIPTION:
This is an open-label study intended to evaluate the relative bioavailability of 4 Probuphine implants versus 16mg QD sublingual buprenorphine, as determined by plasma BPN AUC(0-24), during 24 hours at steady state. This study will also provide open-label safety and tolerability data in patients treated with Probuphine.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily provide written informed consent prior to the conduct of any study related procedures
* Male or female, 18-75 years of age
* Meet the DSM-IV criteria for current opioid dependence
* Females of childbearing potential and fertile males must use a reliable means of contraception

Exclusion Criteria:

* Current diagnosis of Acquired Immune Deficiency Syndrome (AIDS)
* Received treatment for opioid dependence (e.g., methadone, BPN) within the previous 90 days
* Current diagnosis of chronic pain requiring opioids for treatment
* Candidates for only short term opioid treatment or opioid detoxification therapy
* Pregnant or lactating females
* Previous hypersensitivity or allergy to BPN or EVA-containing substances or naloxone
* Current use of agents metabolized through Cytochrome P450 3A4 (CYP 3A4) such as azole antifungals (e.g., ketoconazole), macrolide antibiotics (e.g., erythromycin), and protease inhibitors (e.g., ritonavir, indinavir, and saquinavir)
* Current history of coagulopathy, and/or anti-coagulant therapy (such as warfarin)
* Meet the DSM-IV criteria for current dependence on any other psychoactive substances other than opioids or nicotine (e.g., alcohol, sedatives)
* Current use of benzodiazepines other than physician prescribed use
* Significant medical or psychiatric symptoms, cognitive impairment, or other factors which in the opinion of the Investigators would preclude compliance with the protocol, patient safety, adequate cooperation in the study, or obtaining informed consent
* Concurrent medical conditions (such as severe respiratory insufficiency) that may prevent the patient from safely participating in study; and/or any pending legal action that could prohibit participation and/or compliance in study
* Participated in a clinical study within the previous 8 weeks
* Previous participation in a Probuphine clinical trial
* Presence of aspartate aminotransferase (AST) levels greater than or equal to 3 X upper limit of normal and/or alanine aminotransferase (ALT) levels greater than or equal to 3 X upper limit of normal and/or total bilirubin greater than or equal to 1.5 X upper limit of normal and/or creatinine greater than or equal to 1.5 X upper limit of normal
* Clinically significant low platelet count with current history of coagulopathy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2008-09; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Plasma BPN AUC(0-24)during 24 hours at steady state. | Day -1, Day -2 and Week 4

SECONDARY OUTCOMES:
Plasma BPN and NorBPN Cmax | week 4
Time to maximum plasma BPN and NorBPN concentration (tmax) | Day -2, Day -1 and Day 1
Plasma BPN and NorBPN AUC(0-24) during 24 hours at steady state | week 4
Change in plasma BPN concentration | 24 weeks
Number of subjects with adverse events as a measure of safety and tolerability | approx. 11 weeks (due to study termination)
  Adverse events that occurred after the signing of informed consent until 14 days after study drug treatment has been discontinued, or AEs designated as possibly-related to study drug and Serious AEs until resolution or stabilization, were followed.

CONTACTS AND LOCATIONS:
Locations (1):
- Segal Institute For Clinical Research, Fort Lauderdale, Florida, United States

REFERENCES:
- See also: Related Info — http://www.titanpharm.com